CLINICAL TRIAL: NCT05294341
Title: Pilot Study Examining the Pharmacokinetics of 0.35mg Norethindrone vs 5mg Norethindrone Acetate
Brief Title: Metabolism of 0.35mg Norethindrone vs 5mg Norethindrone Acetate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Horvath, MD, MSHP, Assistant Professor of Obstetrics and Gynecology, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19587
Record Dates: First submitted 2022-03-01; First posted 2022-03-24 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Contraception
Keywords: pharmacokinetics; pilot study
MeSH Terms: interventions — Norethindrone Acetate; Norethindrone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug 1 (Active Comparator): Half of the subjects will be assigned 0.35mg norethindrone pills daily for 7 days.
  The other half of the subjects will be 5mg norethindrone acetate pills daily for 7 days.
  Interventions: Drug: Norethindrone Acetate 5 MG; Drug: Norethindrone 0.35 MG
- Drug 2 (Active Comparator): Half of the subjects will be assigned 5mg norethindrone acetate pills daily for 7 days.
  The other half of the subjects will be 0.35mg norethindrone pills daily for 7 days.
  Interventions: Drug: Norethindrone Acetate 5 MG; Drug: Norethindrone 0.35 MG

INTERVENTIONS:
Drug: Norethindrone Acetate 5 MG — As specified in arm design
Drug: Norethindrone 0.35 MG — As specified in arm design

SUMMARY:
0.35mg norethindrone, also known as progesterone only pills, are routinely prescribed as immediate postpartum oral contraception. Norethindrone acetate is prescribed for gynecologic indications, but has never been studied as an efficacious form of contraception. This is a pilot crossover study examining the pharmacokinetics of norethindrone, the metabolically active component of both drugs, in participants taking 5mg norethindrone and 0.35mg norethindrone acetate.

DETAILED DESCRIPTION:
Progesterone only pills are utilized as immediate postpartum contraception. Though it is demonstrated to be safe as contraception, it is known to be less efficacious than other forms of progestin-only contraception, such as DMPA injections, etonogestrel implant insertion, or progestin-containing intrauterine devices. This is largely secondary to its short half-life. Norethindrone acetate is known to have a longer half-life than norethindrone. Though it is widely used in various gynecologic settings, it has never been studied as a contraceptive option. The metabolically active component of norethindrone is norethindrone itself. This study aims to confirm that amounts of norethindrone are comparable or greater in participants taking 5mg of norethindrone acetate vs taking 0.35mg norethindrone, thereby demonstrating the ability to prescribe 5mg norethindrone acetate as a safe and efficacious form of contraception.

This is a pilot crossover study that will study the pharmacokinetics of norethindrone vs norethindrone acetate. 6 subjects will be a part of this study. Three will be assigned to 0.35mg norethindrone as the initial drug and three will be assigned to 5 mg norethindrone acetate as the initial drug. Starting on day 1-3 of the menstrual cycle, participants will start taking Drug 1 at 7:30am every morning for Days 1-7. At 8am Day 1-7 participants will present to the the Clinical Research Laboratory at Milton S. Hershey Medical Center for an 8am blood draw to examine serum norethindrone levels. On Day 8 participants will stop taking the medication. On Day 8 subjects will present to the Clinical Research Lab and will have an IV placed. Participants will get a pregnancy test to rule-out pregnancy and then hourly blood draws from 8am to 4pm to examine serum norethindrone levels. Participants will also fill out a Symptom Diary detailing side effects and overall satisfaction with the drug.

Additionally, on Days 1 and 21, participants will have serum levels drawn to evaluate levels of luteinizing hormone, follicle stimulating hormone, estradiol, and progesterone levels.

Participants will undergo a one month washout. For Cycle 2, the alternate drug will be administered and monitored in the process as detailed above.

The serum samples will be collected in batches, will be spun down and stored in a -4 degree freezer. Levels of norethindrone in serum samples will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-55yo
2. Menstrual length cycles 24-34 days
3. Previously on non-hormonal forms of contraception
4. Ability to follow-up routinely

Exclusion Criteria:

1. Current pregnancy
2. History of anovulatory cycles
3. Irregular cycles (PCOS)
4. On hormonal-based contraception or HRT in past 3 months
5. Infertility or active hormonal treatment of infertility in past 3 months
6. Hx of hysterectomy
7. Postpartum <3 months
8. H/o liver disease, kidney disease, breast cancer, venous thromboembolism
9. Unwilling to use barrier contraception or abstinence
10. Inability to follow-up routinely

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 5mg Norethindrone Acetate, Then 0.35mg Norethindrone: Participants first received 5mg norethindrone acetate first, then 0.35mg norethindrone. They self-administered 5mg norethindrone acetate between 6-8am on days 1-7 of the study. They then proceeded to get phlebotomy drawn one hour after taking 5mg norethindrone acetate. They then stopped taking 5mg norethindrone acetate day 8, and presented for hourly phlebotomy hourly, for 8 hours.
  They they underwent a 1 month washout. Participants then received 0.35mg norethindrone. They self-administered 0.35mg norethindrone between 6-8am on days 1-7 of the study. They then proceeded to get phlebotomy drawn one hour after taking 0.35mg norethindrone. They then stopped taking 0.35mg norethindrone day 8, and presented for hourly phlebotomy hourly, for 8 hours.
- 0.35mg Norethindrone, Then 5mg Norethindrone Acetate: Participants first received 0.35mg norethindrone acetate first, then 5mg norethindrone acetate. They self-administered 0.35mg norethindrone between 6-8am on days 1-7 of the study. They then proceeded to get phlebotomy drawn one hour after taking 0.35mg norethindrone. They then stopped taking 0.35mg norethindrone day 8, and presented for hourly phlebotomy hourly, for 8 hours.
  They they underwent a 1 month washout. Participants then received 5mg norethindrone acetate. They self-administered 5mg norethindrone acetate between 6-8am on days 1-7 of the study. They then proceeded to get phlebotomy drawn one hour after taking 5mg norethindrone acetate. They then stopped taking 5mg norethindrone acetate day 8, and presented for hourly phlebotomy hourly, for 8 hours.
Period: Overall Study
Arm/Group | 5mg Norethindrone Acetate, Then 0.35mg Norethindrone | 0.35mg Norethindrone, Then 5mg Norethindrone Acetate
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence 1: Sequence 1: 0.35mg norethindrone first, then 5mg norethindrone acetate
- Sequence 2: Sequence 2: 5mg norethindrone acetate first, then 0.35mg norethindrone
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (2) | 32 (2) | 30 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
Regular menstrual cycles, not on hormonal contraception [Count of Participants; unit: Participants] | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Serum Concentration of Norethindrone
Description: The change in serum concentration of norethindrone in individuals taking 0.35mg norethindrone and 5mg norethindrone acetate will be assessed daily over one week of medication use. Norethindrone levels are then averaged across all subjects teaching each medication in each sequence for days 1-7.
Time Frame: Day 1-7
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- 5mg Norethindrone Acetate: These norethindrone levels were obtained via daily plasma samples on days 1-7 when subjects were assigned 5mg norethindrone acetate.
- 0.35mg Norethindrone: These norethindrone levels were obtained via daily plasma samples on days 1-7 when subjects were assigned 0.35mg norethindrone.
Arm/Group | 5mg Norethindrone Acetate | 0.35mg Norethindrone
Number analyzed (Participants) | 6 | 6
ng/ml
  Day 1 | 15.69 (8.6) | 2.28 (1.878562984)
  Day 2 | 13.56 (8.695089814) | 2.50 (2.02)
  Day 3 | 13.96 (9.767023293) | 2.28 (1.28)
  Day 4 | 16.56 (9.173183846) | 2.42 (1.08)
  Day 5 | 11.82 (9.173183846) | 2.22 (1.65)
  Day 6 | 18.92 (8.652213867) | 2.82 (1.65)
  Day 7 | 11.30 (6.505930925) | 2.22 (1.30)

2. Secondary Outcome: Day 8 Norethindrone Levels
Description: The change in serum concentration of norethindrone in individuals taking 0.35mg norethindrone and 5mg norethindrone acetate will be assessed hourly for 8 hours in the absence of exposure to either medication. This is represented as a rate of decline.
Time Frame: Hourly for eight hours on Day 8
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 5mg Norethindrone Acetate; 0.35mg Norethindrone: Norethindrone levels were obtained via hourly plasma samples on day 8 for 8 hours when subjects were assigned 5mg norethindrone acetate.
Arm/Group | 5mg Norethindrone Acetate | 0.35mg Norethindrone
Number analyzed (Participants) | 6 | 6
ng/mL
  Hour 0 | 1.54 (0.583608153) | 0.14729 (0.07215209)
  Hour 1 | 1.17 (0.389190923) | 0.129893333 (0.079030195)
  Hour 2 | 1.31 (0.451133779) | 0.149843333 (0.071421545)
  Hour 3 | 1.29 (0.535815038) | 0.112873333 (0.076)
  Hour 4 | 1.13 (0.480888744) | 0.11 (0.084)
  Hour 5 | 1.04 (0.367513739) | 0.11041 (0.11041)
  Hour 6 | 0.99 (0.38615963) | 0.096743333 (0.067140596)
  Hour 7 | 1.0 (0.433300735) | 0.090736667 (0.0645776)
  Hour 8 | 1.03 (0.463022482) | 0.089563333 (0.063464118)

3. Secondary Outcome: Differences of Serum Levels of Estradiol, Luteinizing Hormone (LH), Follicle Stimulating Hormone (FSH), and Progesterone
Description: The serum levels of estradiol, LH, FSH, and progesterone will be compared in individuals taking 0.35mg norethindrone and 5mg norethindrone acetate at study start and on Day 21
Time Frame: Day 1 and Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 5mg Norethindrone Acetate: LH, FSH, estradiol, progesterone levels were obtained on days 1 and 21 when subjects were assigned 5mg norethindrone acetate. Serum levels of each hormone were averaged across all subjects on each day.
- 0.35mg Norethindrone: LH, FSH, progesterone levels were obtained on days 1 and 21 when subjects were assigned 0.35mg norethindrone. Serum levels of each hormone were averaged across all subjects on each day.
Arm/Group | 5mg Norethindrone Acetate | 0.35mg Norethindrone
Number analyzed (Participants) | 6 | 6
ng/mL
  Estradiol Day 1 | 34.7 (9.44) | 33.5 (7.8)
  Estradiol Day 21 | 147 (176) | 139 (56.45)
  Progesterone Day 1 | 0.45 (0.19) | 0.44 (0.16)
  Progesterone Day 21 | 0.95 (0.97) | 11.6 (3.72)
  LH Day 1 | 6.73 (1.56) | 7.4 (1.4)
  LH Day 21 | 11.8 (9.7) | 6.65 (5.37)
  FSH Day 1 | 8.73 (3.5) | 8.53 (3.2)
  FSH Day 21 | 6.7 (3.1) | 2.75 (0.3)

ADVERSE EVENTS:
Time Frame: Approximately 3 months
Groups:
- 5mg Norethindrone: Adverse events were evaluated in all subjects when they were assigned 5mg norethindrone acetate
- 0.35mg Norethindrone: Adverse events were evaluated in all subjects when they were assigned 0.35mg norethindrone
Arm/Group | 5mg Norethindrone | 0.35mg Norethindrone
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT05294341/Prot_SAP_003.pdf
  • Informed Consent Form (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT05294341/ICF_001.pdf